CLINICAL TRIAL: NCT06524193
Title: Comparing Face-to-face Group Voice Therapy to Telepractice Group Voice Therapy for Muscle Tension Dysphonia: A Non-inferiority Randomized Controlled Trial
Brief Title: RCT Face-to-face Group Voice Therapy vs Telepractice Group Voice Therapy for Muscle Tension Dysphonia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Thomas Law, Assistant Professor & Deputy Chief of Division, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CREC Ref. No.: 2022.378; Project No. CUHK 14106422 (Other Grant/Funding Number: General Research Fund)
Record Dates: First submitted 2024-05-21; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Voice Disorders; Muscle Tension Dysphonia; Aphonia
Keywords: Voice Disorders; Muscle Tension Dysphonia; Group Therapy; Telepractice; Service Delivery Model of Voice Therapy; Voice Therapy; Randomised controlled trail
MeSH Terms: conditions — Voice Disorders; Aphonia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of this study, where the mode of therapy received is obvious to the patients, double blinding is not possible. However, single blinding will be adopted in this study. Although all outcome measures data collection will be conducted by the study team clinicians, the coding of data, video and audio analysis will be conducted anonymously by research staff members who do not have knowledge about the group assignments and the time-point of the data collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telepractice group voice therapy (Experimental): Voice therapy delivered in group basis via telepractice.
  Interventions: Behavioral: Telepractice group voice therapy
- Face-to-face group voice therapy (Active Comparator): Voice therapy that will be delivered in group basis in-person with patients.
  Interventions: Behavioral: Face-to-face group voice therapy

INTERVENTIONS:
Behavioral: Telepractice group voice therapy — * Voice therapy delivered in group basis via telepractice.
  * The voice therapy program will include both indirect and direct voice therapy, in accordance with the current best practice recommendations. Indirect voice therapy will include information counselling on voice production and disorder and vocal hygiene. Direct voice therapy will adopt the resonant voice therapy approach and also head and neck relaxation exercises, which has shown to be effective for muscle tension dysphonia.
  Arms: Telepractice group voice therapy
Behavioral: Face-to-face group voice therapy — * Voice therapy that will be delivered in group basis in-person with patients.
  * The voice therapy program will include both indirect and direct voice therapy, in accordance with the current best practice recommendations. Indirect voice therapy will include information counselling on voice production and disorder and vocal hygiene. Direct voice therapy will adopt the resonant voice therapy approach and also head and neck relaxation exercises, which has shown to be effective for muscle tension dysphonia.
  Arms: Face-to-face group voice therapy

SUMMARY:
The goal of this clinical trial is to compare face-to-face group voice therapy to telepractice group voice therapy for muscle tension dysphonia (MTD). The main questions it aims to answer are:

* The effectiveness of telepractice voice therapy for MTD using a randomized controlled trial study design.
* The effectiveness of telepractice group voice therapy using a randomized controlled trial study design.

Participants will receive telepractice group voice therapy or face-to-face group voice therapy. Researchers will compare telepractice group voice therapy to face-to-face group voice therapy for patients with MTD to see if it has the same effectiveness.

DETAILED DESCRIPTION:
STUDY OBJECTIVES

1. Primary Objectives

   1. To evaluate the effectiveness of telepractice voice therapy for MTD using a randomized controlled trial study design.
   2. To evaluate the effectiveness of telepractice group voice therapy using a randomized controlled trial study design.
2. Secondary Objectives

   1. To compare therapy dropout rate and treatment schedule adherence rate of the two modes of group voice therapy (comparing telepractice to face-to-face mode).
   2. To conduct cost-analysis to compare the health-service cost and patient-related cost of the telepractice and face-to-face group voice therapy.
   3. To further investigate the role of group climate in contributing to treatment outcome in group voice therapy.

BACKGROUND

1. Muscle tension dysphonia

   1. Types and prevalence Muscle tension dysphonia (MTD) is a type of voice disorder that is characterized by excessive paralaryngeal musculature tension during phonation. There are two types of MTD, primary and secondary. Primary MTD is associated with the absence of organic vocal fold pathology, whereas secondary MTD is associated with the presence of organic vocal fold pathology.

      MTD is a prevalent voice disorder which constitutes up to 40% of the total voice disorder caseload. In Hong Kong, a study by our team also showed that MTD was highly prevalent in every four primary school teachers, one would have some degree of MTD.
   2. Cause, risk factors and impact The cause of MTD is multifactorial, including incorrect voicing techniques, phonotraumatic behaviours (such as yelling, screaming, and prolonged voice use), psychological and personality factors, compensation of an underlying disease (such as organic vocal fold pathology, reflux disorder, respiratory tract infection). Risk factors for MTD include female sex, lower education level and people in vocations with high vocal demands.

   MTD not only disrupts a person's voice quality but also their efficiency to produce voice for communication leading to impaired psychological wellbeing, reduced job performance, and economic loss due to workplace absenteeism.
2. Voice therapy is the treatment for MTD

   The current gold standard treatment for primary MTD is behavioural voice therapy delivered by speech-language pathologists. For secondary MTD, behavioural voice therapy is recommended for those with vocal fold nodules. However, for other benign vocal fold pathologies, such as vocal polyps, cysts and granuloma, may require phonosurgery as their primary treatment modality.
   1. Disadvantages of the traditional individual voice therapy Traditionally, voice therapy is delivered on a one-to-one basis, where speech-language pathologists provide therapy to the patients individually. However, our team and other researchers reported that individual voice therapy incurs a higher cost, increases the waiting time for therapy and has a higher therapy dropout rate. In particular, poor therapy attendance rate not only jeopardizes clinical outcomes but also wastes healthcare resources.
   2. Group voice therapy is effective and has many benefits Recent studies, including a treatment study by our team, showed that voice therapy when delivered in groups are as effective as individual therapy. In addition to offsetting the disadvantages of individual therapy, our study and other researchers also showed that group voice therapy provided psychosocial support to the group members and facilitated better therapy skills acquisition through group learning. Furthermore, our team also showed that, when a positive group climate is developed, it could lead to better treatment outcome and could reduce therapy dropout rate. Group climate is the patient's perception of therapeutic relationship in the group therapy environment.
3. Delivering voice therapy via telepractice

   In addition to the individual and group model of service delivery, voice therapy has also been extended into telepractice. Our team was among the first to introduce and provide preliminary evidence to support the use of telepractice in voice therapy for patients with MTD.
   1. The reason for telepractice voice therapy Telepractice was initially applied to voice therapy with the aim to reduce service access barriers due to traveling requirements, work commitments and access to experienced clinicians and patient mobility. However, due to the arrival of COVID-19 pandemic, social distancing policies and lockdowns have caused an abrupt disruption of all in-person voice therapy programs.

      This has left thousands of patients worldwide without any treatment and hence has prolonged and aggravated the negative impact on their professional careers and emotional well-being. Even for those who can attend in-person voice therapy, they are likely to be required to wear masks to mitigate COVID-19 transmission risk. It is important to understand that mask wearing can affect a person's voice quality and production. As such, the treatment effect would unavoidably be impacted.
   2. The urgent need for evidence to support telepractice voice therapy. However, after these initial preliminary findings, no further research on telepractice voice therapy for MTD was conducted. Not until the arrival of COVID-19 pandemic since 2019, researchers and clinicians see the urgency to substantiate the efficacy of telepractice due to its increasing demands and utilization across the globe. Nevertheless, with the limited studies available, researchers were only able to publish recommendation guidelines to guide clinicians in providing voice therapy via telepractice.
4. A lack of study on telepractice voice therapy for MTD and on group therapy

Following the preliminary studies on telepractice voice therapy published in 2015, only two additional studies were found in the literature on telepractice voice therapy. Although both studies showed that the effectiveness of telepractice voice therapy is comparable to face-to-face therapy, they were provided on an individual basis and on different clinical populations. One study focused on the elderly population with various types of voice disorders and the other study focused on voice prevention for those who are at risk at developing voice disorder.

To date, there are no high-quality clinical trials investigating the effectiveness of telepractice voice therapy for patients with MTD, especially when delivered in a group model.

ELIGIBILITY:
Inclusion Criteria:

* Above or equal to 18 years of age;
* Diagnosis of primary MTD or secondary MTD where voice therapy is the primary mode of treatment, such as vocal fold nodules;
* Chinese-speaking subjects only.

Exclusion Criteria:

* Dysphonia of neurogenic or psychogenic origin;
* Secondary muscle tension dysphonia in which voice therapy is not the primary treatment modality, such as vocal polyp, vocal cyst, granuloma, papilloma;
* Low computer literacy or without social or family support for telepractice;
* Patients who are not capable of making own consent;
* Patients who are receiving other modalities of treatment which is not part of this current study, such as traditional Chinese medicine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in patient-related outcome measure | Baseline (before the intervention), 2 weeks follow-up, 3 months follow-up, 6 months follow-up
  The Chinese Voice-Handicap Index (VHI-30) is a reliable patient-related outcome measure. It provides an overall measurement of a person's vocal function and how it influences on a person's everyday functioning and experience. VHI-30 has 30 items. Each item is rated on a scale from with 0 as never, 1 as almost never, 2 as sometimes, 3 as almost always, and 4 as always.
  Statistical analysis: Two-way repeated measures of ANOVA to compare between group performance. To allow for non-inferiority analysis, the 95% confidence interval of the difference in VHI scores between the two groups will be calculated. The upper limit of the 95% CI will be used to determine whether the difference between group is within the non-inferiority margin.
Change in laryngeal imaging | Baseline (before the intervention), 2 weeks follow-up, 3 months follow-up, 6 months follow-up
  Videostroboscopy will be conducted to identify anatomical and physiological outcomes. These include presence of laryngeal pathology, laryngeal physiological patterns. Two experienced laryngologists blinded to the patient's information will rate the video recordings.
  Statistical analysis: Reliability measures will be applied using intraclass correlation for both intra and interrater reliability. Perceptual evaluation of voice will be conducted using two-way repeated measures of ANOVA. Non-inferiority analysis will be also conducted.
Change in perceptual evaluation of voice | Baseline (before the intervention), 2 weeks follow-up, 3 months follow-up, 6 months follow-up
  Patients' voice quality will be assessed using the Cantonese Perceptual Evaluation of Voice scale (Thomas Law, Lee, Lam, van Hasselt, & Tong, 2013). Two experienced speech-language pathologists blinded to the patient's information will rate the audio recordings.
  Statistical analysis: Reliability measures will be applied using intraclass correlation for both intra and interrater reliability. Perceptual evaluation of voice will be conducted using two-way repeated measures of ANOVA. Non-inferiority analysis will be also conducted.
Change in acoustic voice analysis | Baseline (before the intervention), 2 weeks follow-up, 3 months follow-up, 6 months follow-up
  The Computerized Speech Lab system will be used to measure parameters including jitter, shimmer, and noise-to-harmonic ratio and cepstral peak prominence.
  Statistical analysis: Acoustic analysis will be conducted using two-way repeated measures of ANOVA. Non-inferiority analysis will be also conducted.
Change in aerodynamic measures | Baseline (before the intervention), 2 weeks follow-up, 3 months follow-up, 6 months follow-up
  Maximum phonation time will be measured.
  Statistical analysis: Aerodynamic measure will be conducted using two-way repeated measures of ANOVA. Non-inferiority analysis will be also conducted.

SECONDARY OUTCOMES:
Therapy dropout rate and treatment schedule adherence rate | Immediately after the intervention
  This will be measured by comparing the proportion of patient dropout and non-adherence to treatment schedule in both modes of treatment.
  Statistical analysis will be conducted using the Z-test.
Cost analysis | Immediately after the intervention
  This will follow the cost analysis approach suggested by Burns and colleagues. Cost domains including human resource cost, patient cost and equipment cost.
  Statistical analysis will be conducted using the t-test.
Group climate | Immediately after the intervention
  The group climate questionnaire will be used to measure the therapeutic relationship at the final session of each therapy group.
  Statistical analysis: the contribution of group climate to treatment outcome will be measured using correlation analysis and one-way repeated ANOVA.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Law, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Division of Speech Therapy, Dept of Otorhinolaryngology , Head and Neck Surgery, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abrahamsson M, Millgard M, Havstam C, Tuomi L. Effects of Voice Therapy: A Comparison Between Individual and Group Therapy. J Voice. 2018 Jul;32(4):437-442. doi: 10.1016/j.jvoice.2017.06.008. Epub 2017 Jul 18. PMID 28732752
- [Background] Altman KW, Atkinson C, Lazarus C. Current and emerging concepts in muscle tension dysphonia: a 30-month review. J Voice. 2005 Jun;19(2):261-7. doi: 10.1016/j.jvoice.2004.03.007. PMID 15907440
- [Background] Becker DR, Gillespie AI. In the Zoom Where It Happened: Telepractice and the Voice Clinic in 2020. Semin Speech Lang. 2021 Jan;42(1):64-72. doi: 10.1055/s-0040-1722750. Epub 2021 Feb 17. PMID 33596605
- [Background] Burns CL, Kularatna S, Ward EC, Hill AJ, Byrnes J, Kenny LM. Cost analysis of a speech pathology synchronous telepractice service for patients with head and neck cancer. Head Neck. 2017 Dec;39(12):2470-2480. doi: 10.1002/hed.24916. Epub 2017 Sep 30. PMID 28963804
- [Background] Cantarella G, Torretta S, Ferruta S, Ciabatta A, Manfredi C, Pignataro L, Dejonckere P. Multidimensional Assessment of the Effectiveness of Group Voice Therapy. J Voice. 2017 Nov;31(6):714-721. doi: 10.1016/j.jvoice.2017.02.004. Epub 2017 Mar 1. PMID 28259606
- [Background] Castillo-Allendes A, Contreras-Ruston F, Cantor-Cutiva LC, Codino J, Guzman M, Malebran C, Manzano C, Pavez A, Vaiano T, Wilder F, Behlau M. Voice Therapy in the Context of the COVID-19 Pandemic: Guidelines for Clinical Practice. J Voice. 2021 Sep;35(5):717-727. doi: 10.1016/j.jvoice.2020.08.001. Epub 2020 Aug 7. PMID 32878736
- [Background] DeVore EK, Carroll TL, Rosner B, Shin JJ. Can voice disorders matter as much as life-threatening comorbidities to patients' general health? Laryngoscope. 2020 Oct;130(10):2405-2411. doi: 10.1002/lary.28417. Epub 2019 Dec 3. PMID 31794064
- [Background] Eastwood C, Madill C, Mccabe P. The behavioural treatment of muscle tension voice disorders: A systematic review. Int J Speech Lang Pathol. 2015 Jun;17(3):287-303. doi: 10.3109/17549507.2015.1024169. Epub 2015 May 8. PMID 25953458
- [Background] Lin FC, Chien HY, Chen SH, Kao YC, Cheng PW, Wang CT. Voice Therapy for Benign Voice Disorders in the Elderly: A Randomized Controlled Trial Comparing Telepractice and Conventional Face-to-Face Therapy. J Speech Lang Hear Res. 2020 Jul 20;63(7):2132-2140. doi: 10.1044/2020_JSLHR-19-00364. Epub 2020 Jun 24. PMID 32579859
- [Background] Fu S, Theodoros DG, Ward EC. Delivery of Intensive Voice Therapy for Vocal Fold Nodules Via Telepractice: A Pilot Feasibility and Efficacy Study. J Voice. 2015 Nov;29(6):696-706. doi: 10.1016/j.jvoice.2014.12.003. Epub 2015 Feb 26. PMID 25726070
- [Background] Fu S, Theodoros DG, Ward EC. Intensive versus traditional voice therapy for vocal nodules: perceptual, physiological, acoustic and aerodynamic changes. J Voice. 2015 Mar;29(2):260.e31-44. doi: 10.1016/j.jvoice.2014.06.005. Epub 2014 Oct 12. PMID 25311594
- [Background] Grillo EU. Building a Successful Voice Telepractice Program. Perspect ASHA Spec Interest Groups. 2019 Feb;4(1):100-110. doi: 10.1044/2018_PERS-SIG3-2018-0014. PMID 31544152
- [Background] Grillo EU. A Nonrandomized Trial for Student Teachers of an In-Person and Telepractice Global Voice Prevention and Therapy Model With Estill Voice Training Assessed by the VoiceEvalU8 App. Am J Speech Lang Pathol. 2021 Mar 26;30(2):566-583. doi: 10.1044/2020_AJSLP-20-00200. Epub 2021 Feb 1. PMID 33524262
- [Background] Hapner E, Portone-Maira C, Johns MM 3rd. A study of voice therapy dropout. J Voice. 2009 May;23(3):337-40. doi: 10.1016/j.jvoice.2007.10.009. PMID 18674882
- [Background] Iwarsson J. Facilitating behavioral learning and habit change in voice therapy--theoretic premises and practical strategies. Logoped Phoniatr Vocol. 2015 Dec;40(4):179-86. doi: 10.3109/14015439.2014.936498. Epub 2014 Jul 23. PMID 25054888
- [Background] Knickerbocker K, Bryan C, Ziegler A. Phonogenic Voice Problems among Speech-Language Pathologists in Synchronous Telepractice: An Overview and Recommendations. Semin Speech Lang. 2021 Jan;42(1):73-84. doi: 10.1055/s-0040-1722754. Epub 2021 Feb 17. PMID 33596606
- [Background] Lam PK, Chan KM, Ho WK, Kwong E, Yiu EM, Wei WI. Cross-cultural adaptation and validation of the Chinese Voice Handicap Index-10. Laryngoscope. 2006 Jul;116(7):1192-8. doi: 10.1097/01.mlg.0000224539.41003.93. PMID 16826059
- [Background] Law T, Lee KY, Ho FN, Vlantis AC, van Hasselt AC, Tong MC. The effectiveness of group voice therapy: a group climate perspective. J Voice. 2012 Mar;26(2):e41-8. doi: 10.1016/j.jvoice.2010.12.003. Epub 2011 May 7. PMID 21550777
- [Background] Ng E, Law T, Tang EC, Ho FN, Tong MC, Lee KY. The Cutoff Point and Diagnostic Accuracy of the Voice Handicap Index in Cantonese-Speaking Population. J Voice. 2021 Mar;35(2):163-168. doi: 10.1016/j.jvoice.2020.09.021. Epub 2020 Oct 9. PMID 33046276
- [Background] Nguyen DD, McCabe P, Thomas D, Purcell A, Doble M, Novakovic D, Chacon A, Madill C. Acoustic voice characteristics with and without wearing a facemask. Sci Rep. 2021 Mar 11;11(1):5651. doi: 10.1038/s41598-021-85130-8. PMID 33707509
- [Background] Ohlsson AC, Dotevall H, Gustavsson I, Hofling K, Wahle U, Osterlind C. Voice Therapy Outcome-A Randomized Clinical Trial Comparing Individual Voice Therapy, Therapy in Group, and Controls Without Therapy. J Voice. 2020 Mar;34(2):303.e17-303.e26. doi: 10.1016/j.jvoice.2018.08.023. Epub 2018 Oct 19. PMID 30344071
- [Background] Portone C, Johns MM 3rd, Hapner ER. A review of patient adherence to the recommendation for voice therapy. J Voice. 2008 Mar;22(2):192-6. doi: 10.1016/j.jvoice.2006.09.009. Epub 2007 Jun 15. PMID 17572065
- [Background] Rangarathnam B, McCullough GH, Pickett H, Zraick RI, Tulunay-Ugur O, McCullough KC. Telepractice Versus In-Person Delivery of Voice Therapy for Primary Muscle Tension Dysphonia. Am J Speech Lang Pathol. 2015 Aug;24(3):386-99. doi: 10.1044/2015_AJSLP-14-0017. PMID 25836732
- [Background] Roy N, Barkmeier-Kraemer J, Eadie T, Sivasankar MP, Mehta D, Paul D, Hillman R. Evidence-based clinical voice assessment: a systematic review. Am J Speech Lang Pathol. 2013 May;22(2):212-26. doi: 10.1044/1058-0360(2012/12-0014). Epub 2012 Nov 26. PMID 23184134
- [Background] Roy N. Functional dysphonia. Curr Opin Otolaryngol Head Neck Surg. 2003 Jun;11(3):144-8. doi: 10.1097/00020840-200306000-00002. PMID 12923352
- [Background] Ruotsalainen J, Sellman J, Lehto L, Verbeek J. Systematic review of the treatment of functional dysphonia and prevention of voice disorders. Otolaryngol Head Neck Surg. 2008 May;138(5):557-65. doi: 10.1016/j.otohns.2008.01.014. PMID 18439458
- [Background] Ruotsalainen JH, Sellman J, Lehto L, Jauhiainen M, Verbeek JH. Interventions for treating functional dysphonia in adults. Cochrane Database Syst Rev. 2007 Jul 18;(3):CD006373. doi: 10.1002/14651858.CD006373.pub2. PMID 17636842
- [Background] Simberg S, Sala E, Tuomainen J, Sellman J, Ronnemaa AM. The effectiveness of group therapy for students with mild voice disorders: a controlled clinical trial. J Voice. 2006 Mar;20(1):97-109. doi: 10.1016/j.jvoice.2005.01.002. Epub 2005 Jun 16. PMID 15963687
- [Background] Speyer R. Effects of voice therapy: a systematic review. J Voice. 2008 Sep;22(5):565-80. doi: 10.1016/j.jvoice.2006.10.005. Epub 2007 May 16. PMID 17509828
- [Background] Trajano FMP, Almeida LNA, de Alencar SAL, Braga JEF, Almeida AA. Group Voice Therapy Reduces Anxiety in Patients With Dysphonia. J Voice. 2020 Sep;34(5):702-708. doi: 10.1016/j.jvoice.2019.03.003. Epub 2019 Apr 9. PMID 30979532
- [Background] Van Houtte E, Claeys S, Wuyts F, Van Lierde K. The impact of voice disorders among teachers: vocal complaints, treatment-seeking behavior, knowledge of vocal care, and voice-related absenteeism. J Voice. 2011 Sep;25(5):570-5. doi: 10.1016/j.jvoice.2010.04.008. Epub 2010 Jul 15. PMID 20634042
- [Background] Van Houtte E, Van Lierde K, Claeys S. Pathophysiology and treatment of muscle tension dysphonia: a review of the current knowledge. J Voice. 2011 Mar;25(2):202-7. doi: 10.1016/j.jvoice.2009.10.009. Epub 2010 Apr 18. PMID 20400263
- [Background] Van Houtte E, Van Lierde K, D'Haeseleer E, Claeys S. The prevalence of laryngeal pathology in a treatment-seeking population with dysphonia. Laryngoscope. 2010 Feb;120(2):306-12. doi: 10.1002/lary.20696. PMID 19957345
- [Background] Verdolini K, Ramig LO. Review: occupational risks for voice problems. Logoped Phoniatr Vocol. 2001;26(1):37-46. PMID 11432413
- [Background] Hall N, Boisvert M, Steele R. Telepractice in the assessment and treatment of individuals with aphasia: a systematic review. Int J Telerehabil. 2013 Jun 11;5(1):27-38. doi: 10.5195/ijt.2013.6119. eCollection 2013 Spring. PMID 25945211
- [Background] White A. Management of benign vocal fold lesions: current perspectives on the role for voice therapy. Curr Opin Otolaryngol Head Neck Surg. 2019 Jun;27(3):185-190. doi: 10.1097/MOO.0000000000000536. PMID 30893134
- [Background] Yiu EM, Lo MC, Barrett EA. A systematic review of resonant voice therapy. Int J Speech Lang Pathol. 2017 Feb;19(1):17-29. doi: 10.1080/17549507.2016.1226953. Epub 2016 Oct 5. PMID 27705008